CLINICAL TRIAL: NCT00732849
Title: The Impact of the Type and Route of Nutritional Support on Infectious Complications After Upper Gastrointestinal Surgery - A Prospective, Randomized, Clinical Trial.
Brief Title: The Impact of the Type and Route of Nutritional Support on Infectious Complications After Upper Gastrointestinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: 1st Department of General Surgery, Jagiellonian University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: surg nutr
Record Dates: First submitted 2008-08-05; First posted 2008-08-12 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-07

CONDITIONS: Gastrointestinal Surgery
Keywords: immunonutrition; surgical patients; postoperative period
MeSH Terms: interventions — alanylglutamine; fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (No Intervention): Standard Enteral Nutrition - Peptisorb, Nutricia Ltd.
  Interventions: Drug: Reconvan, Dipeptiven, Omegaven
- 2 (No Intervention): Standard Parenteral Nutrition: Aminomel, Lipofundin, Glucose, Cernevit, Tracutil, electrolytes
  Interventions: Drug: Reconvan, Dipeptiven, Omegaven
- 3 (Experimental): Immunomodulating Enteral Nutrition: Reconvan, Fresenius Kabi Poland
  Interventions: Drug: Reconvan, Dipeptiven, Omegaven
- 4 (Experimental): Immunomodulating Parenteral Nutrition: Aminomel, Lipofundin, Glucose, Cernevit, Tracutil, electrolytes + Omegaven (Fresenius Kabi), Dipepitven (Fresenius Kabi)
  Interventions: Drug: Reconvan, Dipeptiven, Omegaven

INTERVENTIONS:
Drug: Reconvan, Dipeptiven, Omegaven — Reconvan (1ml=1 kcal), 30 kcal/kg b.w. Omegaven 1 ml/ kg b.w. Dipeptiven 1 ml/ kg b.w.

SUMMARY:
The study was designed to test the hypothesis that immunonutrition and enteral nutrition would reduce the incidence of infectious complications in a population of malnourished patients following elective upper GI surgery

DETAILED DESCRIPTION:
All patients qualified between June 2002 and December 2007 to total and distal subtotal gastrectomy or pancreaticoduodenectomy were screened for eligibility to participate in the study. Malnutrition was defined by the Nutritional Risk Index (NRI), calculated according to the formula used in the Veterans Administration Cooperative Group trial.{, 1991 #70} Additional eligibility criteria included: age between 18 and 80 years, Karnofsky performance status score of 80 or more, and adequate organ function measured by routine blood tests. Patients without features of malnutrition, as well as those with disseminated tumors, serious comorbidities (American Society of Anesthesiologists risk class of 4 or 5), and renal or liver failure were excluded. The study was designed to test the hypothesis that immunonutrition and enteral nutrition would reduce the incidence of infectious complications in a population of malnourished patients following elective upper GI surgery. Therefore, patients were randomly assigned in a 2×2 factorial design to four groups receiving immunostimulating versus normal diets, and enteral versus intravenous nutritional support. The secondary objective of the study was to evaluate the effect of nutritional intervention on overall morbidity and mortality rates, and the length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years,
* Karnofsky performance status score of 80 or more,
* adequate organ function measured by routine blood tests

Exclusion Criteria:

* patients <18 or > 80
* Karnofsky performance < 50

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2002-06; Primary Completion 2002-09 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Immunonutrition and enteral nutrition would reduce the incidence of infectious complications in a population of malnourished patients | Immunonutrition

SECONDARY OUTCOMES:
To evaluate the effect of nutritional intervention on overall morbidity and mortality rates, and the length of hospital stay | morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw Klek, MD, PhD, Principal Investigator — Jagiellonian University
Locations (1):
- 1st Department of SUegy, Krakow, _30978, Poland